CLINICAL TRIAL: NCT06819150
Title: Effect of Bathing on Physiological Parameters, Skin, Bilirubin and Comfort Levels in Infants Receiving Phototherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Raziye Çelen, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/78_TR
Record Dates: First submitted 2025-01-04; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Phototherapy Skin Rash
Keywords: Phototherapy; Newborn; Bilirubin; Bath; Comfort; Skin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborn bathing (Experimental): The term and preterm infants in the experimental group will have a bathtub bath before starting phototherapy treatment.
  Interventions: Other: Newborn bathing
- Standard of care (No Intervention): No intervention other than routine clinical practices will be applied to the control group.

INTERVENTIONS:
Other: Newborn bathing — The babies in the experimental group will have a bathtub bath before starting phototherapy treatment.
  Arms: Newborn bathing

SUMMARY:
The aim of this study is to determine the effect of bathing on physiological parameters (heart rate, body temperature and oxygen saturation), skin, bilirubin and comfort level in infants receiving phototherapy.

DETAILED DESCRIPTION:
Neonatal jaundice (hyperbilirubinemia) causes a yellowish discolouration of the sclera and skin due to increased levels of bilirubin in the blood. Jaundice develops in 60% of term babies and 80% of premature babies in the first week of life. Currently, the appropriate treatment option for neonatal jaundice is phototherapy. Phototherapy treatment reduces bilirubin concentrations through various photochemical reactions that allow bilirubin to be excreted more easily. However, phototherapy treatment is associated with short-term side effects including transient skin rashes, diarrhoea, hyperthermia and dehydration.

Physiological reasons such as the weak connection between the epidermis and dermis layer in the skin of the newborn, the pH value of the skin being close to neutral or alkaline, and the low melanosome production increase the susceptibility of the newborn to infection and skin damage. Invasive interventions, use of antiseptics, phototherapy and various instruments may disrupt the skin integrity of the newborn. Therefore, all newborns receiving treatment and care in the neonatal intensive care unit are at risk in terms of skin integrity.

In the majority of newborn infants; jaundice develops, which can affect the newborn neurologically, motor and hearing if left untreated,. Phototherapy devices are widely used today for the treatment of jaundice. Phototherapy devices used in the treatment of jaundice have side effects such as skin rashes, diarrhea, dehydration and hyperthermia. In the literature reviewed, results were found that bathing the newborn reduces phototherapy rashes, lowers the bilirubin level and increases the comfort of the newborn. Also in the literature; There are studies showing that one of the most suitable bathing methods for a newborn is bathtub bathing and that bathing with baby shampoo is not harmful to the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Born at 35-41 gestational weeks
* Indirect hyperbilirubinaemia diagnosed at 24 hours of birth or more,
* No health problems,
* Indication for phototherapy treatment
* Stable vital signs
* Whose parents agreed to participate in the study

Exclusion Criteria:

* Newborns with ABO and Rh incompatibility,
* Direct diagnosis of hyperbilirubinaemia,
* Congenital anomaly,
* With skin lesions

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Infant Information Form | First measurement-First day of hospitalization
  The form, prepared by the researchers based on the literature, includes questions containing natal-postnatal information of preterm and term infants (date of birth, gestational week, postnatal age, gender, birth weight, mode of delivery, NICU admission date, initiation time of phototherapy, etc.).
Follow-up form for physiologic parameters - Heart rate | Heart rate will be measured 10 minutes before the intervention (T0), 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after the intervention.
  Heart rate will be measured 10 minutes before the intervention, 30 minutes, 60 minutes and 6 hours after the intervention.
Follow-up form for physiologic parameters -Respiratory rate | Respiratory rate will be measured 10 minutes before the intervention (T0), 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after the intervention.
  Respiratory rate will be measured 10 minutes before the intervention, 30 minutes, 60 minutes and 6 hours after the intervention.
Follow-up form for physiologic parameters- Body temperature | Body temperature will be measured 10 minutes before the intervention (T0), 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after the intervention.
  Body temperature will be measured 10 minutes before the intervention, 30 minutes, 60 minutes and 6 hours after the intervention.
Follow-up form for physiologic parameters- Oxygen saturation | Oxygen saturation will be measured 10 minutes before the intervention (T0), 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after the intervention.
  Oxygen saturation will be measured 10 minutes before the intervention, 30 minutes, 60 minutes and 6 hours after the intervention.
Follow-up form for Skin moisture | Skin moisture will be measured 10 minutes before the intervention (T0), 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after the intervention.
  Skin moisture will be measured using a device (Digital Moisture Monitor for Skin) on the forehead, abdomen, back, arms (right-left) and legs (right-left).
Neonatal Skin Condition Score | Neonatal Skin Condition Assessment Scale, will assess the infants' skin condition 10 minutes before treatment/bath (T0) The infants' skin condition will then be reassessed 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after bath or treatment.
  Neonatal Skin Condition Assessment Scale, will assess the infants' skin condition 10 minutes before treatment/bath (T0) The infants' skin condition will then be reassessed 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after bath or treatment.
Bilirubin level | In the experimental and control groups, the total serum bilirubin levels will be evaluated 10 minutes before treatment/bathing (T0). The bilirubin levels will be measured for the second time at 24 hours after the start of phototherapy treatment (T1).
  In the experimental and control groups, the total serum bilirubin levels will be evaluated 10 minutes before treatment/bathing (T0). The bilirubin levels will be measured for the second time at 24 hours after the start of phototherapy treatment (T1).
The comfort level | The comfort level of the babies in the experimental and control groups will be evaluated 10 minutes before the treatment/bath. The comfort of the babies will be re-evaluated 30 minutes (T1), 60 minutes (T2) and 6 hours (T3) after the bath or treatment.
  The Newborn Comfort Behavior Scale (COMFORTneo) will assess the comfort of the newborn. The scale will evaluate the newborn's calmness/agitation, respiratory response, pain, body movements, facial tension, and muscle tone.The scale is scored between 6-30. As the score obtained from the scale increases, it shows that the newborn is uncomfortable and needs practices that will increase their comfort

CONTACTS AND LOCATIONS:
Overall Officials: Perihan B Çalışkan, MSc student, Principal Investigator — Selcuk University; Raziye Çelen, Asst. Prof., Principal Investigator — Selcuk University
Locations (1):
- Kütahya Şehir Hospital, Kütahya, Merkez, Turkey (Türkiye)